CLINICAL TRIAL: NCT02188043
Title: Relay Model for Recruiting Alcohol Dependent Patients in General Hospitals - A Single-blind Pragmatic Randomised Trial
Brief Title: Project Relay Model for Recruiting Alcohol Dependent Patients in General Hospitals
Acronym: Relay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kjeld Andersen, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RESCueH_Relay
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Alcohol Use Disorder; Alcohol Dependency
Keywords: Alcohol use disorder; Motivational Intervention; Health expenditures; efficacy study
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Relay Model (Other): AUDIT score 8+: Brief Motivational Intervention with alcohol therapist. AUDITscore16+:Brief Motivational Intervention and appointment at Alcohol Treatment Clinic
  -
  Interventions: Behavioral: Relay Model
- Usual Referral Procedure (No Intervention): Hospital staff refer patient to Alcohol Treatment Clinic according to usual procedure

INTERVENTIONS:
Behavioral: Relay Model — The Clinical staff hand out and collect lifestyle - questionnaires to admitted patients, and screen by 10 alcohol questions (AUDIT) , and report score to outpatient Alcohol Clinic.
  Based on the questionnaire that the patient filled out, the Alcohol therapist perform a brief Motivational Intervention on patients with an AUDIT score of 8+, focusing the patients alcohol consumption habits and offer an appointment to patients with an AUDIT score of 16+.
  Arms: Relay Model

SUMMARY:
The purpose of this study is to evaluate the Relay Model helping alcohol dependent patients at a general hospital to start specialized alcohol treatment in order to assess i) efficacy, ii) cost-effectiveness and iii) overall societal cost impacts.

The effect of the Relay Model will be investigated in a single-blind pragmatic randomised controlled trial in which the control group consists of patients referred to treatment by usual procedures.

DETAILED DESCRIPTION:
An increase in individuals with alcohol dependence receiving specialized alcohol treatment will be of major importance for society's response to alcohol problems and its consequences. The Danish population has a large intake of alcohol. Approximately 20% of the adult population are heavy drinkers ( >14/21 drinks/ week (women/men)), 14% are harmful users, and 3% are dependent drinkers. Untreated alcohol use disorders lead to frequent contacts to the health care system associated with considerable human and societal costs. A first approach would be to identify and recruit patients from general hospitals, where the proportion of inpatients with alcohol use disorders range between 16 % and 26%. A referral model to ensure treatment for alcohol dependent patients after discharge is needed.

The main objective of the study is to develop strategies which increase the likelihood that patients report for outpatient alcohol treatment after discharge. It is likely that an optimization of the transfer procedure between hospital and outpatient clinic will lead to that more patients will be engage in psychosocial treatment for their alcohol abuse, which will improve the prognosis, reduce re-admissions and the use of hospital beds and, thus have positive economic consequences. We evaluate the Relay Model in order to assess i) efficacy, ii) cost-effectiveness and iii) overall societal cost impacts.

The target group of the present study is patients suffering from alcohol dependence admitted to a general hospital located in an urban area and a general hospital located in a rural area.

A single-blind pragmatic randomised controlled trial including patients admitted to Hospital. The study group(n=500) receive an Intervention and the control group(n=500) are referred to treatment by usual procedures. All patients complete a lifestyle questionnaire with the Danish self-report version of the Alcohol Use Disorders Identification Test (AUDIT) embedded as a case identification strategy. The patients are informed that an alcohol therapist may contact them and give feedback on their responses.

The completed forms are reviewed daily and an AUDIT score of 8+prompts a call to the Alcohol therapist, who attends the departments on different days randomly drawn by a computer. The RELAY MODEL intervention include a Brief Motivational Intervention. Patients who score AUDIT 16+ are also offered an appointment at the alcohol treatment clinic.

Primary measure is health care expenditures 12 months after discharge, according to the International Classification of Health Accounts, extracted from population registers. The analysis will be repeated on a yearly basis during the following 5 years.

Secondary outcome: The percentage of the target group, who, 30 days after discharge, reports at the alcohol treatment clinics.

A multiple regression model will be used. Since non-treated alcohol disorders generate a high number of societal costs annually for health care, social services, traffic accidents, criminal activities and lost productions we believe the Relay Model to be either cost-neutral or cost-effective, i.e. low net costs compared to effectiveness. We expect to establish evidence that the Relay Model is either cost-neutral or cost-effective, compared to referral by usual procedures.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for a minimum of 24 hours
* Resident within the uptake area of the involved alcohol treatment centres
* Willing to participate in the study
* Cognitive and physical capable

Exclusion Criteria:

* In any alcohol-specific treatment for alcohol dependence
* Psychotic
* Less than 18 years of age
* Hospitalized less than 24 hours
* Resident outside uptake areas
* Not consenting on participation in the study
* Cognitive and physical incapable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
health care expenditures | 12 - 60 months
  Primary measure is Health care expenditures 12 months after discharge, according to the International Classification of Health Accounts, extracted from population registers.

SECONDARY OUTCOMES:
report to alcohol clinic | 30 days
  Secondary outcome is the percentage of the target group, who, 30 days after discharge, reports at the alcohol treatment clinics.

CONTACTS AND LOCATIONS:
Overall Officials: Bent Nielsen, Ph.D, Principal Investigator — bent.nielsen@rsyd.dk
Locations (1):
- RESCueH alcohol Studies, Unit of Clinical Alcohol Research, Psyciatric Research Unit, Clinical Institute, University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Derived] Schwarz AS, Bilberg R, Bjerregaard L, Nielsen B, Sogaard J, Nielsen AS. Relay model for recruiting alcohol dependent patients in general hospitals--a single-blind pragmatic randomized trial. BMC Health Serv Res. 2016 Apr 14;16:132. doi: 10.1186/s12913-016-1376-8. PMID 27080865